CLINICAL TRIAL: NCT07064096
Title: Effects Of Mental Imagery Along With Vestibular Rehabilitation On Young Adults With Vestibular Hypofunction
Acronym: EMI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sulman amjad
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Vestibular Hypofunction
Keywords: VESTIBULAR REHAB WITH MENTAL IMAGERY; BALANCE; VERTIGO AND DIZZINESS

STUDY DESIGN:
Intervention Model Description: Interventional model
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): cawthorne cooksey exercises
  Interventions: Other: cawthorne cooksey exercise
- participatory Group (Experimental): cawthorne cooksey exercises in addition of mental imagery
  Interventions: Other: mental imagery

INTERVENTIONS:
Other: cawthorne cooksey exercise — Cawthorne Cooksey exercises -Start with low to moderate intensity. Cawthorne Cooksey exercise Training Phase1-In bed exerercises:- Eye movements: 1)Up and down 2)Side to side 3)Moving finger away from face -Phase2-Sitting: Eye movements as above. Head movements at firsts low, then quick later with eyes closed -bending forward and backward -turning from side to side. --Shoulder shrugging and circling -Bending forward and picking up objects from the ground - Phase 3 - Standing: -Eye, Head, Shoulder movements -Throwing ball from hand to hand, hand under knee -Switch to sitting to standing and turning around in between. -Phase 4 - Walk: with eyes closed and open: -Across room -Slope and Stairs
  Other Names: cawthorne cooksey exercises
  Arms: Conventional treatment
Other: mental imagery — The mental imagery intervention in this study is a structured, guided cognitive training program designed to enhance the effects of vestibular rehabilitation in young adults with unilateral vestibular hypofunction. Mental imagery (MI) involves the internal visualization and mental rehearsal of physical movements without actual motor output, engaging similar neural pathways as actual execution.
  Arms: participatory Group

SUMMARY:
The objective of the study is to determine the effects of cawthorne cooksey exercises with addition of mental imagery on vertigo,dizziness and balance in young adults with vestibular hypofunctionThe study will be randomized control trial including 2 experimental groups with estimated 22 participants in each group.

DETAILED DESCRIPTION:
The vestibular system detects motion of the head in space and in turn generates reflexes that are crucial for our daily activities, such as stabilizing the visual axis (gaze) and maintaining head and body posture. The vestibular system is comprised of two types of sensors: the two otolith organs (the saccule and utricle), which sense linear acceleration, and the three semicircular canals, which sense angular acceleration in three planes. The receptor cells of the otoliths and semicircular canals send signals through the vestibular nerve fibers to the neural structures that control eye movements, posture, and balance.

Vestibular hypofunction i.e. a unilateral or a bilateral vestibulopathy, is a heterogeneous disorder of the peripheral and/or rarely central vestibular system leading typically to disabling symptoms such as dizziness, imbalance, and/or oscillopsia.

Mental imagery (MI), also known as motor imagery or cognitive rehearsal, is the mental simulation of physical movement without actual execution. MI activates similar brain regions involved in physical movement and has been shown to improve motor performance, balance, and functional outcomes in various populations. However, its application in conjunction with vestibular rehabilitation for individuals with vestibular hypofunction remains underexplored.

This study aims to investigate the combined effect of mental imagery and vestibular rehabilitation exercises on balance, dizziness, and vertigo in young adults diagnosed with vestibular hypofunction. The intervention will involve a structured VR program integrated with guided mental imagery sessions targeting balance and gaze stabilization tasks.

Participants will be randomly assigned to two groups: one receiving only vestibular rehabilitation i.e cawthorne-cooksey exercises and the other receiving both VR and mental imagery training. Outcome measures such as the Dizziness Handicap Inventory (DHI), Mini-BESTest (Mini Balance Evaluation Systems Test and Vertigo Symptom Scale will be used to assess changes pre- and post-intervention.

This research intends to determine whether the addition of mental imagery enhances the efficacy of vestibular rehabilitation in restoring functional balance and reducing dizziness symptoms. The findings could contribute to developing more comprehensive and accessible rehabilitation strategies for managing vestibular disorders in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral vestibular hypofunction
* Head thrust test positive
* Age group 20-40
* DHI score 16 above
* VSS score 11-30

Exclusion Criteria:

* With any other associated neurological disorder that effect vestibular rehabilitation
* Having bilateral vestibular hypofunction
* Patients having any other associated disease that affects balance or cause vertigo other that vestibular

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Vertigo Symptom Scale | 8 week
  The Vertigo Symptom Scale (VSS) is a self-report questionnaire designed to assess the severity and frequency of vertigo-related symptoms over the past month
• Dizziness Handicap Inventory | 8 week
  The Dizziness Handicap Inventory (DHI) is a self-reported questionnaire designed to evaluate the impact of dizziness on a person's daily life, emotional well-being, and functional ability. It is widely used in clinical practice for assessing vestibular dysfunction and tracking progress in rehabilitation. Purpose of DHI is to Measures how dizziness affects daily activities.
Mini-BESTest (Mini Balance Evaluation Systems Test) | 8 week
  The Mini-BESTest is a shortened version of the Balance Evaluation Systems Test (BESTest). It is designed to assess dynamic balance and identify impairments in postural control across different systems. This test is particularly useful for evaluating balance deficits in vestibular disorders

CONTACTS AND LOCATIONS:
Overall Officials: Nadia azhar, MS, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Alnasir Hospital Gujar Khan, Gujar Khān, Punjab Province
  - Riphah International University, Islamabad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu KP, Chan CC, Lee TM, Hui-Chan CW. Mental imagery for promoting relearning for people after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2004 Sep;85(9):1403-8. doi: 10.1016/j.apmr.2003.12.035. PMID 15375808
- [Background] Ellis AW, Schone CG, Vibert D, Caversaccio MD, Mast FW. Cognitive Rehabilitation in Bilateral Vestibular Patients: A Computational Perspective. Front Neurol. 2018 Apr 27;9:286. doi: 10.3389/fneur.2018.00286. eCollection 2018. PMID 29755404
- [Background] van Esch BF, Nobel-Hoff GE, van Benthem PP, van der Zaag-Loonen HJ, Bruintjes TD. Determining vestibular hypofunction: start with the video-head impulse test. Eur Arch Otorhinolaryngol. 2016 Nov;273(11):3733-3739. doi: 10.1007/s00405-016-4055-9. Epub 2016 Apr 25. PMID 27113255